CLINICAL TRIAL: NCT01560754
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center Trial to Assess the Disease-modifying Potential of Transdermal Nicotine in Early Parkinson's Disease in Germany and the USA
Brief Title: Disease-modifying Potential of Transdermal NICotine in Early Parkinson's Disease
Acronym: NIC-PD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: James BOYD MD (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Parkinson Study Group (PSG) (Unknown); International Parkinson Fonds Germany GmbH (Industry); German Parkinson Study Group (GPS) (Other); German Parkinson Society (DPG) (Other); Philipps University Marburg (Other)
Responsible Party: Sponsor-Investigator, James BOYD MD, United States Principal Investigator, University of Vermont
Organization: University of Vermont (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KKS-135
Record Dates: First submitted 2012-03-09; First posted 2012-03-22 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
Keywords: Randomized; Placebo-controlled; Double-blind; Multi-center; Disease-modifying potential; transdermal nicotine
MeSH Terms: conditions — Parkinson Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal nicotine patch (Experimental): Subjects will apply a combination of 7 or 14 mg nicotine transdermal patches until reaching their highest well tolerated dose of 7 to 28 mg/day.
  Interventions: Drug: nicotine transdermal patch
- Transdermal placebo patch (Placebo Comparator): Subjects will apply a combination of 7 or 14 mg placebo transdermal patches until reaching their highest well tolerated dose.
  Interventions: Drug: nicotine transdermal patch

INTERVENTIONS:
Drug: nicotine transdermal patch — Transdermal patches containing 7 or 14 mg nicotine or placebo with subjects titrating up until reaching their highest tolerated dose of 7 to 28mg/day.
  Other Names: Habitrol Transdermal patch (US); Nicotinell Transdermal patch (Germany)

SUMMARY:
The primary objective of this study is to demonstrate that transdermal nicotine treatment retards disease progression as measured by change in total Unified Parkinson's Disease Rating Scale (UPDRS)(part I, II, III)score between baseline and after 52 weeks of study treatment plus two more months wash out (60 weeks).

DETAILED DESCRIPTION:
In order to prove the disease-modifying potential of transdermal nicotine treatment, an explanatory design with a 2 months wash-out phase before endpoint assessment will be performed. The primary objective is to demonstrate superiority measured by the difference between the nicotine arm and the placebo arm in the change in total UPDRS score (part I-III) between baseline and end of month 14 (12 months treatment and 2 months wash-out, see 3.1). The total UPDRS score will be determined by an independent rater, who is not involved in any other study-related procedure (e.g. reporting of adverse events). Change in total UPDRS score is the most widely applied measure in similar clinical trials assessing long-term beneficial effects of drugs. The investigators will also determine whether the slope of the curves for the total UPDRS score in active- and placebo-treated subjects show a tendency to converge over time. For this purpose the UPDRS will be determined three times after placebo/nicotine withdrawal at the end of the study during Visit 7,8, and 9 (i.e. four times including Visit 6).

Approximately 250 subjects will be screened at 25-30 centers in Germany and the USA. The recruitment period will be 18 months. In the screening phase, subjects will be evaluated for eligibility for enrolment into the treatment phase. The investigators expect that screening of 250 subjects will result in 160 eligible subjects who will be randomly assigned 1:1 to treatment with either transdermal nicotine or transdermal placebo patch.

The treatment phase consists of a titration period (16 weeks, to find the highest dosage tolerated by the subject with a target of 28 mg) and a maintenance period (week 17 to week 52 with the highest tolerated dosage of nicotine).

The treatment phase will be followed by an 8 week wash-out phase (3 weeks down titration and 5 weeks run out).

Dose adjustments are permitted for adverse events and have to be documented thoroughly.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Capability and willingness to comply with the study related procedures
3. Age >/= 30 y
4. Usage of effective contraception (see below) in fertile pre-menopausal female participants (from inclusion until end of wash out) Acceptable forms of effective contraception include established use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception (condom or occlusive cap /diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository or male / female sterilization / or true abstinence.
5. Diagnosis of PD according to the UK Brain Bank Diagnostic Criteria
6. Early PD subjects within 18 months of diagnosis
7. Hoehn and Yahr stage ≤ 2
8. Patients not receiving or needing dopamine agonist or levodopa therapy presently or for the next year
9. Stable treatment (>2 months) with MAO-B inhibitor (selegiline up to 10 mg/d or rasagiline up to 1 mg/d) allowable

Exclusion Criteria:

1. Clinical signs indicating a Parkinson syndrome other than idiopathic PD e.g.:

   * Supranuclear gaze palsy
   * Signs of frontal dementia
   * History of repeated strokes with stepwise progression of Parkinsonian features
   * History of repeated head injury or history of definite encephalitis
   * Cerebellar signs
   * Early severe autonomic involvement
   * Babinski's sign
2. History of exposure to or current treatment with neuroleptic drugs or anticraving substances
3. History of nicotine use within five years of the baseline visit
4. Previous history of allergic response to nicotine application or any of the patch excipients (see protocol sec. 10.2)
5. Previous history of allergic response to transdermal patches
6. Pre-existing dermatological disorder that could disturb transdermal patch application in the opinion of the investigator (e.g. generalized / systemic or local neurodermatitis, psoriasis, chronic dermatitis, urticaria, etc.)
7. Previous treatment with antiparkinsonian drugs (e.g. levodopa, dopamine agonists, etc.) other than MAO-B inhibitors
8. History of unstable or serious cardiovascular diseases

   * Unstable or worsening angina pectoris,
   * History of recent myocardial infarction or cardiac failure (NYHA from II to IV), myocardial insufficiency
   * History at inclusion of serious cardiac arrhythmia,
   * History of recent stroke or occlusive peripheral vascular disease, vasospasm
9. History of structural brain disease, cerebrovascular diseases
10. History of severe uncontrolled arterial hypertension
11. History of severe pulmonary disease (asthma, COPD)
12. History of auto-immune disease
13. History of Hyperthyroidism
14. History of Pheochromocytoma
15. History of seizures / epilepsy
16. History of amyosthenia / myasthenia gravis, pseudo-myasthenic syndrome
17. Dementia defined as Mini Mental State Examination (MMSE) score ≤ 24
18. Moderate depression (BDI-II score >24)
19. Suicide or suicide ideation
20. History or presence of specific psychiatric disorders, acute psychosis, hallucinations, pathologic gambling, alcohol or substance abuse
21. Patients under treatment with dihydropyridines (e.g. nifedipine, nicardipine, amlodipine)
22. History of uncontrolled diabetes
23. History of recent gastroduodenal ulcer (< 3 months) or presence of severe (acute and chronic) gastritis
24. History of known hepatobiliary or renal insufficiency
25. Pregnancy or lactation period
26. Simultaneous participation or previous participation within 60 days before screening in another clinical drug or medical device study. Other Trials that do not affect the NIC-PD Study (NIT, health economics evaluations, questionnaires, genetic studies) could be allowed, but have to be approved and documented by the steering committee

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is calculated as the difference between the nicotine arm and the placebo arm in the change in total UPDRS I-III score between baseline and 60 weeks (14 months) (52 weeks treatment plus 8 weeks wash-out). | From Baseline to week 60
  The primary objective is to demonstrate superiority measured by the difference between the nicotine arm and the placebo arm in the change in total UPDRS score (part I-III) between baseline and end of month 14 (12 months treatment and 2 months wash-out

SECONDARY OUTCOMES:
The change in total UPDRS I-III score between baseline and 52 weeks (12 months) | Baseline to 52 weeks
Parkinson's Disease Questionaire - 8(PDQ-8) that is calculated as the change between baseline and 60 weeks | Baseline and week 60
The frequency of adverse events will be analyzed | Baseline through week 60
The 'time to initiation of a symptomatic treatment' is calculated from the date of randomization to the date that a subject initiates symptomatic therapy | Baseline to initiation of symptomatic therapy, this timeframe will vary from subject to subject based on duration of disease and how well their PD is currently being managed
Determine whether the slope of the curves for the total UPDRS score in active- and placebo-treated subjects show a tendency to converge over time | Baseline to week 52 and week 60
Parkinson's Disease Questionnaire - 8 (PDQ-8), a patient completed questionaire, calculated as the change between baseline and week 52 | Baseline and week 52
Scales for Outcomes of Parkinson's disease - Cognition (SCOPA-COG), is calculated as the change between baseline and week 52 | Baseline and week 52
Beck Depression Inventory - II (BDI-II) that is calculated as the change between baseline and week 52 | Baseline and week 52
Parkinson's Disease Sleep Scale (PDSS) that is calculated as the change between baseline and week 52 | baseline and week 52
SCOPA-COG that is calculated as the change between baseline and 60 weeks | Baseline and week 60
BDI-II that is calculated as the change between baseline and 60 weeks | Baseline and Week 60
PDSS that is calculated as the change between baseline and week 60 | Baseline and Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Oertel, MD, Principal Investigator — Philipps-University Marburg, Germany / Global and German Principal Investigator; James Boyd, MD, Principal Investigator — University of Vermont / United States Principal Investigator
Locations (24):
- United States (9):
  - University of Southern California, Los Angeles, California
  - The Parkinsons Institute, Sunnyvale, California
  - Pacific Health Research & Education Institute, Honolulu, Hawaii
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Struthers Parkinson'S Center, Golden Valley, Minnesota
  - Feinstein Institute For Medical Research, North Shore-Lij Health System, Manhasset, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont
- Germany (15):
  - Universitatsklinikum Giessen U. Marburg GmbH, Standort Marburg, Marburg
  - Charite Campus Virchow Klinikum, Berlin
  - Klinikum Bremerhaven, Bremerhaven
  - Universitaetsklinikum CarlGustav Carus, Dresden
  - Neurologische Klinik der, Dusseldorf, Düsseldorf
  - Neurologische Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Klinikum Hanau GmbH, Hanau
  - Universitaetsklinikum des Saarlandes, Homburg/Saar
  - Paracelsus-Elena-Klinik Kassel, Kassel
  - Universitaetsklinikum Schlewsig-Holstein, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Otto-von-Guericke-Universitat, Magdeburg
  - Klinikum rechts der Isar, München
  - Universitaetsklinikum Tubingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Oertel WH, Muller HH, Unger MM, Schade-Brittinger C, Balthasar K, Articus K, Brinkman M, Venuto CS, Tracik F, Eberling J, Eggert KM, Kamp C, Kieburtz K, Boyd JT. Transdermal Nicotine Treatment and Progression of Early Parkinson's Disease. NEJM Evid. 2023 Sep;2(9):EVIDoa2200311. doi: 10.1056/EVIDoa2200311. Epub 2023 Aug 22. PMID 38320207